CLINICAL TRIAL: NCT06834906
Title: Usability User Testing of the Easy-EyeFM AI Platform
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tsinghua University (Other)
Collaborators: First Hospital of Tsinghua University (Other); Beijing Tsinghua Changgeng Hospital (Other); Augenarzt-Praxisgemeinschaft Gutblick AG (Unknown); Sankara Nethralaya (Other); Department of Medical Services Ministry of Public Health of Thailand (Other Government); Moorfields Eye Hospital NHS Foundation Trust (Other); Pomeranian Hospitals (Unknown); Shanghai Health and Medical Center (Unknown); Hong Kong Eye Hospital (Other); Royal Victoria Eye and Ear Hospital (Other Government); Hanyang University Guri Hospitall (Unknown); Alshifa Trust Eye Hospital (Unknown); Korle-Bu Teaching Hospital, Accra, Ghana (Other); Nippon Medical School Tama Nagayama Hospital (Unknown)
Responsible Party: Principal Investigator, Tien Yin Wong, Professor, Tsinghua University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Easy-EyeFM
Record Dates: First submitted 2025-02-09; First posted 2025-02-19 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-01

CONDITIONS: Ocular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Experimental)
  Interventions: Diagnostic Test: EasyEyeFM-AutoML-AI-platform test
- group B (Experimental)
  Interventions: Diagnostic Test: AutoML-EasyEyeFM-AI-platform test

INTERVENTIONS:
Diagnostic Test: EasyEyeFM-AutoML-AI-platform test — AI platforms using
  Arms: group A
Diagnostic Test: AutoML-EasyEyeFM-AI-platform test — AI-platform using
  Arms: group B

SUMMARY:
Easy-EyeFM is a code-free artificial intelligence platform designed for ophthalmologists to provide diagnostic and treatment recommendations and help doctors develop customized diagnostic models.

This project aims to evaluate the usability and user-friendliness of the Easy-EyeFM platform for physicians. The study will gather feedback from medical professionals to evaluate the intuitiveness and effectiveness of the platform in supporting model customization and medical image analysis tasks.

Subjects will participate in the trial of the Easy-EyeFM platform and the comparison with the existing commercial platform (AutoML) at the appointed time. The researchers will inform subjects of relevant precautions and assist them to read the user manual before the test. Subjects will complete model customization and picture diagnosis within the prescribed test time, and according to the test results, Score the human-computer interaction experience of the AI platform, fill in the questionnaire, and finally complete the evaluation content.

ELIGIBILITY:
Inclusion Criteria:

* Medical students or doctors
* Have enough time to participate in this program, about 1 hour continuous assessment
* Agree to sign the informed consent form

Exclusion Criteria:

* Poor computer and mobile phone use and reading ability
* Poor language expression or dialect category is not included in the speech recognition function of the platform

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-01-26 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | 1 day
  Minimum Value: 0 Maximum Value: 100 Higher scores indicate a better outcome, meaning higher system usability.

SECONDARY OUTCOMES:
Usage Time | 1 day
Users Assistance Requests Times | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Tien Yin Wong, Principal Investigator — Tsinghua University
Locations (1):
- Tsinghua University, Beijing, China

IPD SHARING:
Plan to Share IPD: No